CLINICAL TRIAL: NCT02516267
Title: The Importance of Evaluation of Platelet Aggregability in the Release of Coronary Artery Bypass Grafting in Patients With Acute Coronary Syndrome With Dual Antiplatelet Therapy.
Brief Title: Evaluation of Platelet Aggregability in the Release of CABG in Patients With ACS With DAPT.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Carlos Alberto Kenji Nakashima, Medical Doctor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Multiplate CABG
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Bleeding
Keywords: platelet aggregability; acute coronary syndrome; coronary artery bypass graft
MeSH Terms: conditions — Hemorrhage; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): Patients who will discontinue inhibitor-ADP for 5 days before surgery, and must be operated on the first working day after completing the 5 days without the drug. This group will have its aggregability evaluated by platelet function testing (Multiplate ADP®) immediately before the transport to the operating room.
- Intervention Group (Active Comparator): Patients will be evaluated by platelet function testing (Multiplate ADP®) daily until the value obtained> 46 AU, when they will be immediately released to CABG, to be held on the first working day after release.
  Interventions: Device: Multiplate ADP®

INTERVENTIONS:
Device: Multiplate ADP® — Patients will be evaluated by platelet function testing (Multiplate ADP®) daily until the value obtained> 46 AU, when they will be immediately released to CABG
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to assess platelet aggregability by a "point of care" device (Multiplate®) to decrease the release time for coronary artery bypass graft (CABG ) in patients with acute coronary syndrome (ACS) in use of dual antiplatelet therapy.

DETAILED DESCRIPTION:
This open, prospective, randomized study will be included patients with acute coronary syndrome (ACS) and coronary artery bypass graft (CABG) indication in use of double platelet aggregation (aspirin and inhibitor of ADP). The groups to be analyzed will be:

1. Control group: It is composed of patients who will discontinue inhibitor of ADP for 5 days before surgery, and must be operated on the first working day after completing the 5 days without the drug. This group will have aggregability evaluated by platelet function testing (Multiplate®) immediately before the transport to the operating room.
2. Intervention group: It is composed of patients who will be evaluated by platelet function testing (Multiplate®) daily until the value obtained> 46 AU, when they will be immediately released to CABG, to be held on the first working day after release.

All patients included, after the explanations and signing the informed consent, will initially undergo preoperative examinations as institutional routine. In the immediate period (24 hours) after CABG will be collected on all results of tests to which the patient is submitted in accordance with the institutional routines, and the volume of chest tube bleeding and need for blood transfusions. Clinical data "MACE" will be collected throughout the patient's hospital stay.

ELIGIBILITY:
Inclusion Criteria:

1. Age> 18 years;
2. Hospitalization for ACS defined as:

   - Symptoms ischemic unstable pattern, occurring at rest or upon exertion within 72 hours of an unscheduled hospitalization, related to presumed or proven coronary artery, and at least one of the following:
   * elevated cardiac biomarkers (troponin I or CK-MB mass) above the 99th percentile.
   * Changes in resting electrocardiogram compatible with ischemia or infarction and further evidence of obstructive coronary artery disease:

   the resting ECG compatible with ischemia or infarction in at least one of the criteria below:
   * ST segment depression of new or presumably new> 0.5 mm in 2 sequential leads.
   * The new ST-segment elevation or presumed new J point in two contínguas leads with value> 0.2mV in men or> 0.15mV in women in V2-V3 and / or> 0.1mV in other leads or new left bundle branch block or presumably again.
   * T wave inversion new or presumably new> 1mm in leads with a broad R wave in two contiguous leads.
   * New pathological Q wave or presumably new> 30 ms duration and> 1mm deep in 2 contiguous leads or> 20 ms or QS complex in V2 and V3.
   * Peaked new R Wave> 40 ms in V1 and V2, R / S> 1 in V1 with positive T wave in the absence of consistent driving change.
   * Additional evidence of coronary artery disease in at least one of the criteria below:
   * Evidence of myocardial ischemia or new or presumably new in imaging with perfusion.
   * Contractility Change in new or presumably new wall.
   * Coronary angiography with obstruction> 70% in epicardial coronary artery.
3. Use of dual antiplatelet therapy (ASA associated with P2Y12 receptor inhibitor);
4. An indication of CABG.
5. Agreement to sign the Informed Consent (IC);

Exclusion criteria:

1. anemia (hematocrit <30%).
2. Thrombocytopenia (<100,000 / mm³).
3. Coagulopathy (history of bleeding diathesis or use of oral anticoagulants).
4. Chronic renal failure dialysis or creatinine clearance <30 ml / min / m2 (estimated by MDRD formula).
5. Active liver disease.
6. combined valvuloplasty or valve replacement surgery ..
7. Angioplasty with stent for less than 30 days or with drug-eluting stents for less than one year.
8. Use of fibrinolytic specific fibrin not less than 48 hours or specific fibrin less than 24 hours of randomization;
9. Any medical condition that in the investigator's opinion present significant risk to the patient or interfere with the interpretation of the safety and efficacy;
10. Patients who are taking part in another clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2015-07; Primary Completion 2015-07 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Bleeding by chest tubes in 24 hours postoperative. | 24 hours postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carlos Nicolau, Cardiology, Study Chair — Heart Institute (HC/FMUSP)
Locations (1):
- Carlos Alberto Kenji Nakashima, São Paulo, Brazil

REFERENCES:
- [Derived] Nakashima CAK, Dallan LAO, Lisboa LAF, Jatene FB, Hajjar LA, Soeiro AM, Furtado RHM, Dalcoquio TF, Baracioli LM, Lima FG, Giraldez RRCV, Silva BA, Costa MSS, Strunz CMC, Dallan LRP, Barbosa CJDG, Britto FAB, Farkouh ME, Gurbel PA, Nicolau JC. Platelet Reactivity in Patients With Acute Coronary Syndromes Awaiting Surgical Revascularization. J Am Coll Cardiol. 2021 Mar 16;77(10):1277-1286. doi: 10.1016/j.jacc.2021.01.015. PMID 33706868